CLINICAL TRIAL: NCT01206036
Title: Phase I/II Study With Temsirolimus Versus no add-on in Patients With Castration Resistant Prostate Cancer (CRPC) Receiving First-line Docetaxel Chemotherapy
Brief Title: CESAR Study in Prostate Cancer With Temsirolimus Added to Standard Docetaxel Therapy (CEPTAS)
Acronym: CEPTAS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Central European Society for Anticancer Drug Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-II-007; 2010-018370-21 (EudraCT Number)
Record Dates: First submitted 2010-08-17; First posted 2010-09-21 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Prostatic Neoplasms
Keywords: castration; prostate cancer; castration resistant prostate cancer; PSA; Docetaxel; Temsirolimus; disease progression free survival; DPFS; dose escalation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Docetaxel — DL 1: Docetaxel 60mg/m^2, Temsirolimus 15mg. DL 2: Docetaxel 60mg/m^2, Temsirolimus 25mg. DL 3: Docetaxel 75mg/m^2, Temsirolimus 25mg. One cycle is defined as a 3 week period (21 days) where docetaxel is given on day 1, and temsirolimus on days 1, 8 and 15.
  Other Names: Taxotere
Drug: Temsirolimus — DL 1: Docetaxel 60mg/m^2, Temsirolimus 15mg. DL 2: Docetaxel 60mg/m^2, Temsirolimus 25mg. DL 3: Docetaxel 75mg/m^2, Temsirolimus 25mg. One cycle is defined as a 3 week period (21 days) where docetaxel is given on day 1, and temsirolimus on days 1, 8 and 15.
  Other Names: Torisel

SUMMARY:
In this Phase I study safety of the combination of Docetaxel and Temsirolimus needs to be shown before the study can be expanded into a Phase II study to examine the activity of a safe combination of Temsirolimus and Docetaxel in a comparison with Docetaxel alone.

DETAILED DESCRIPTION:
The purpose of this Phase I study is to evaluate feasibility of dose levels DL1, DL2 and DL3 (which are combinations of Temsirolimus and Docetaxel) and defining a recommended dose (RD) for the Phase II part using these dose levels in a dose escalating scheme.

Secondary objectives are the collection of safety data on the dose levels used in this part.

ELIGIBILITY:
Inclusion Criteria Phase I Part:

* Adult males ≥18 years of age.
* Patients with CRPC defined as confirmed rise of PSA levels after orchiectomy or LHRH agonist based therapy.
* Progressive disease, defined as PSA progression by confirmed rising PSA levels.
* PSA at time of study entry ≥2ng/ml within 1 week prior to treatment (according to Scher 2008).
* Bone metastasis and/or lymph node and/or visceral organ metastases allowed. Measurable and non measurable disease allowed.
* Performance status (PS) 0-1 ECOG.
* Signed written informed consent.
* White blood cell count (WBC) ≥4x10^9/L with neutrophils ≥1.5x10^9/L, platelet count ≥100x10^9/L, hemoglobin ≥9g/dL.
* Total bilirubin <=2 x upper limit of normal.
* AST and ALT <=2.5 x upper limit of normal, or <=5 x upper limit of normal in case of liver metastases.
* Serum creatinine <=1.5 x upper limit of normal or creatinine clearance > 60 ml/min.
* Androgen ablation will have to be continued. Antiandrogens such as bicalutamide will have to be discontinued at least 4 weeks prior to the start of study treatment.

Exclusion Criteria Phase I Part:

* Clinically symptomatic brain or meningeal metastasis.
* Receiving known strong CYP3A4 isoenzyme inhibitors and/or inducers.
* Any investigational drug within the 30 days before inclusion.
* Not recovered from prior biopsy, surgery, traumatic injury, and/or radiation therapy, as judged by the investigator.
* Nonhealing wound or ulcer.
* Grade ≥ 3 hemorrhage within the past month.
* Any condition / concomitant disease not allowing chemotherapy with docetaxel, prednisone and temsirolimus in the discretion of the treating physician, like: Renal insufficiency requiring dialyses; congestive heart failure or uncontrolled angina pectoris; prior myocardial infarction within 6 months of start of chemotherapy; uncontrolled severe hypertension (failure of diastolic blood pressure to fall below 90 mm Hg despite the use of ≥ 3 anti-hypertensive drugs) or arrhythmias; instable diabetes mellitus, ulceration from diabetes mellitus or other conditions not allowing high dose corticosteroids; effusions in pericardium, pleura or abdomen symptomatic and in need of being punctured.
* Known hypersensitivity to any of the components in the temsirolimus infusion or other medical reasons for not being able to receive adequate premedication (antihistamine agents).
* Legal incapacity or limited legal capacity
* Medical or psychological conditions that would not permit the patient to
* complete the study or sign informed consent.

Inclusion Criteria Phase II Part, Chemotherapy Period:

* Adult males ≥ 18 years of age.
* Patients with CRPC defined as confirmed rise of PSA levels after orchiectomy or LHRH agonist based therapy
* Progressive disease, defined as PSA progression by confirmed rising PSA levels
* PSA at time of study entry ≥ 2ng/ml within 1 week prior to treatment (according to Scher 2008).
* Bone metastasis and/or lymph node and/or visceral organ metastases allowed. Measurable and non measurable disease allowed.
* Performance status (PS) 0-1 ECOG.
* Signed written informed consent.
* White blood cell count (WBC) ≥4x10^9/L with neutrophils ≥1.5x10^9/L, platelet count ≥100x10^9/L, hemoglobin ≥9g/dL.
* Total bilirubin <= 2 x upper limit of normal.
* AST and ALT <=2.5 x upper limit of normal, or <=5 x upper limit of normal in case of liver metastases.
* Serum creatinine <=1.5 x upper limit of normal or creatinine clearance >60 ml/min.
* Androgen ablation will have to be continued. Antiandrogens such as bicalutamide will have to be discontinued at least 4 weeks prior to the start of study treatment.

Exclusion Criteria Phase II Part, Chemotherapy Period:

* Prior Chemotherapy.
* Clinically symptomatic brain or meningeal metastasis.
* Receiving known strong CYP3A4 isoenzyme inhibitors and/or inducers.
* Any investigational drug within the 30 days before inclusion.
* Not recovered from prior biopsy, surgery, traumatic injury, and/or radiation therapy, as judged by the investigator.
* Nonhealing wound or ulcer.
* Grade ≥ 3 hemorrhage within the past month.
* Any condition / concomitant disease not allowing chemotherapy with docetaxel, prednisone and temsirolimus in the discretion of the treating physician, like: Renal insufficiency requiring dialyses; congestive heart failure or uncontrolled angina pectoris; prior myocardial infarction within 6 months of start of chemotherapy; uncontrolled severe hypertension (failure of diastolic blood pressure to fall below 90 mm Hg despite the use of ≥ 3 anti-hypertensive drugs) or arrhythmias; instable diabetes mellitus, ulceration from diabetes mellitus or other conditions not allowing high dose corticosteroids; effusions in pericardium, pleura or abdomen symptomatic and in need of being punctured.
* Known hypersensitivity to any of the components in the temsirolimus infusion or other medical reasons for not being able to receive adequate premedication (antihistamine agents).
* Legal incapacity or limited legal capacity.
* Medical or psychological conditions that would not permit the patient to complete the study or sign informed consent.

Inclusion Criteria Phase II Part, Maintenance Period:

* Completed 8 cycles (up to 26 weeks) treatment in Arm A
* White blood cell count (WBC) ≥4x10^9/L with neutrophils ≥1.5x10^9/L, platelet count ≥100x10^9/L, hemoglobin ≥9g/dL.
* Total bilirubin <=2 x upper limit of normal.
* AST and ALT <=2.5 x upper limit of normal, or <=5 x upper limit of normal in case of liver metastases.
* Serum creatinine <=1.5 x upper limit of normal or creatinine clearance >60 ml/min.
* General condition sufficient to allow therapy with temsirolimus.
* Signed Informed Consent.

Exclusion Criteria Phase II Part, Maintenance Period:

* Disease Progression in the first 8 cycles (up to 26 weeks).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-07; Primary Completion 2014-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
recommended dose | 10 months
  Phase I Part: Primary endpoint is the Recommended Dose (RD) for the Phase II Part chosen between the three DLs based on the dose escalation scheme.
disease progression-free survival | 24 months
  Phase II Part: Primary endpoint is to evaluate the activity of the addition of Temsirolimus to standard treatment on the disease progression-free survival (DPFS Chemotherapy) in patients with castration resistant prostate cancer receiving first-line Docetaxel chemotherapy.

SECONDARY OUTCOMES:
safety as defined as occurence of treatment related adverse events | 10 months
  Phase I Part: Secondary endpoint is the collection of safety data on the dose levels used in this part.
overall response | 24 months
  Phase II Part: Responses of measurable disease (RECIST 1.1 criteria) including the overall response rate (RR, CFR+PR) and the disease control rate (PR+CR+SD). In addition to the overall response rate RR, the trial will also evaluate the number of responders based on PSA evaluation only (RR-PSA) and the number of responders based on RECIST evaluation only (RR-RECIST) among those who are evaluable by that criterion, respectively. RR is only evaluated for the chemotherapy part of the Phase II part of the trial.
1-year Disease-Progression Free Survival Rate | 24 months
  Phase II Part: 1-year Disease-Progression Free Survival Rate (DPFS-1yR); defined as the quotient defined exactly in the same way as DPFS-6mR with the landmark time point equal to 1 year, +/- 4 weeks for assessment one year after randomization.
DPFS time | 24 months
  Phase II Part: DPFS time measured as failure time between 1st randomization and disease progression or death whatever occurred first. Patients lost-to follow-up, dropping out (e.g. when withdrawing consent) or patients surviving progression free at the end-of-study time point are treated as censored cases.
TTP-PSA | 24 months
  Phase II Part: Time to PSA progression (TTP-PSA) measured from randomization until PSA progression as defined in Scher et al. "Decline from baseline: record time from start of therapy to first PSA increase that is ≥ 25% and ≥ 2 ng/mL above the nadir, and which is confirmed by a second value 3 or more weeks later (ie, a confirmed rising trend)†"
toxicity based on treatment-related toxicities using CTCAE v4.0 | 24 months
  Phase II Part: Evaluation of toxicity using CTCAE v4.0
PSA | 24 months
  Phase II Part: Proportion of patients with drop of PSA of > 30% in the evaluation period compared to baseline compared to baseline.
quality of life | 24 months
  Phase II Part: Quality of life using the EORTC questionnaire
overall survival | 24 months
  Phase II Part: overall survival (OS) measured from randomization until death or lost to follow up (censored survival time)
Frequency of medication for pain | 24 months
  Phase II Part: Frequency of medication for pain

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Morant, MD, Study Chair — Tumor-und Brustzentrum ZeTuP, St. Gallen, Switzerland
Locations (2):
- Germany (2):
  - CESAR Study Center, Essen
  - CESAR Study Center, Freiburg im Breisgau

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: web page of CESAR (Central European Society for Anticancer Drug Research-EEIG) — http://www.cesar.or.at